CLINICAL TRIAL: NCT01595932
Title: Efficacy and Tolerability of α-galactosidase in Treating Gas-related Symptoms in Children. A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Efficacy and Tolerability of α-galactosidase in Treating Gas-related Symptoms in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Giovanni Di Nardo, MD, Azienda Policlinico Umberto I
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: α-galactosidase
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Gas Pain Related Intake
Keywords: irritable bowel syndrome (IBS); bloating; abdominal distension; flatulence; α-Galactosidase
MeSH Terms: conditions — Irritable Bowel Syndrome; Flatulence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- α-galactosidase (Experimental)
  Interventions: Dietary Supplement: α-galactosidase

INTERVENTIONS:
Dietary Supplement: α-galactosidase — Treatment was administered at the beginning of each meal (3 times a day) for 2 weeks:
  children < 20kg: 4 drops;
  children > 20kg and < 40kg: 8 drops;
  children > 40kg: 1 tablet.
  Other Names: Sinaire
  Arms: α-galactosidase
Dietary Supplement: Placebo — Treatment was administered at the beginning of each meal (3 times a day) for 2 weeks:
  children < 20kg: 4 drops;
  children > 20kg and < 40kg: 8 drops;
  children > 40kg: 1 tablet.
  Arms: placebo

SUMMARY:
The aim of this study was to evaluate the efficacy and tolerability of α-galactosidase in pediatric patients with predominant gas-related symptoms.

DETAILED DESCRIPTION:
Most patients with functional gastrointestinal disorders complain of gas-related symptoms which can negatively affect quality of life, even in pediatric age.

Dietary and life-style changes, administration of simethicone, activated charcoal and probiotics may reduce intestinal gas but often results are unsatisfactory.

Literature shows that α-galactosidase is effective to reduce gas production and related symptoms in adults.

ELIGIBILITY:
Inclusion Criteria:

* pediatric out-patients with gas-related disturbances at least once per week over the last 12 weeks.

Exclusion Criteria:

* suspected episodes of hypersensitivity or allergy;
* chronic organic disorders (by clinical history, physical examination, laboratory tests);
* use of drug affecting the GI motility during the previous 4 weeks;
* inability of the parent to comprehend the full nature and purpose of the study and unwillingness to co-operate with the Investigator.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Efficacy | 5 weeks of observation
  Global distress associated with gas-related symptoms (bloating, flatulance, abdominal distension and abdominal spasm): data collected by parents or patients on a daily diary chart, 3 time/daily by using a validated visual score scale (Faces Pain Scale-Revised).

SECONDARY OUTCOMES:
Clinical tolerability | treatment: 2 weeks
  Recording of all Adverse Events (AEs) occurred during the 2 weeks of treatment
Efficacy | 5 weeks of observation (baseline: 1 week; treatment: 2 weeks; follow-up: 2 weeks)
  Frequency and intensity (6 point scale: 0=absent; 5=very severe)of bloating, flatulance, visible distension, spasms.
  Data were collected by parents or patients on a daily diary chart.
Efficacy | 5 weeks of observation (baseline: 1 week; treatment: 2 weeks; follow-up: 2 weeks)
  Physician's overall evaluation: 4 point scale (from completed/marked improvement to worse).

REFERENCES:
- [Derived] Di Nardo G, Oliva S, Ferrari F, Mallardo S, Barbara G, Cremon C, Aloi M, Cucchiara S. Efficacy and tolerability of alpha-galactosidase in treating gas-related symptoms in children: a randomized, double-blind, placebo controlled trial. BMC Gastroenterol. 2013 Sep 24;13:142. doi: 10.1186/1471-230X-13-142. PMID 24063420